CLINICAL TRIAL: NCT07300683
Title: Fratricide-Resistant Autologous Chimeric Antigen Receptor T Cells Targeting CCR9 for the Treatment of T Cell Acute Lymphoblastic Leukaemia/ Lymphoma
Brief Title: Anti-CCR9 CAR T Cells for T Cell Leukaemia/Lymphoma
Acronym: FRACTALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Great Ormond Street Hospital Charity (Unknown); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/150854; 2022-003497-23 (EudraCT Number); ISRCTN15341827 (Other: ISRCTN)
Record Dates: First submitted 2025-09-15; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: T Cell Acute Lymphoblastic Leukemia; T Cell Lymphoblastic Lymphoma
Keywords: FRACTALL; Fratricide-Resistant; CCR9; CAR T cells
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, non-randomised, open-label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) for patients with high-risk, relapsed/refractory (r/r) T-ALL/T-LBL.
  The trial will have 2 cohorts: Adult (≥18 years old) and Paediatric (<18 years old).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous anti-CCR9 CAR T cells (Experimental): Patients will receive autologous anti-CCR9 CAR T cells intravenously.
  Interventions: Biological: CARCCR9 T cells

INTERVENTIONS:
Biological: CARCCR9 T cells — Anti-CCR9 CAR T cells

SUMMARY:
The goal of this clinical trial is to learn if anti-CCR9 CAR T cells (which will be made using the patient's own blood cells) are safe and which dose should be used in children and adults with T cell leukaemia and lymphoma.

Participants will:

* have T cells collected from their blood and these T cells will be used to make the CAR-T cells in a specialized laboratory.
* be admitted at the hospital a week before the CAR T cells infusion to receive a short course of chemotherapy drugs which prepare the body to receive the CAR T cells.
* be given the CAR T cells into their vein.
* stay in the hospital for a minimum of 2 weeks to be closely monitored
* following discharge, participants will come to the clinic for check-ups (approximately 12 visits in the first two years)
* during screening, treatment and follow up visits, participants will have physical examination, collection of blood samples and bone marrow biopsies and/or imaging tests (CT/PET-CT scans) depending on their type of T-cell cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsed or refractory T-ALL/T-LBL following at least one (≥18 years old) or two (<18 years old) standard prior lines of combination cytotoxic therapy
* CCR9-positive disease as assessed by flow cytometry
* T-LBL patients only: Patients must have measurable disease
* Agreement to have a pregnancy test, use adequate contraception (if applicable)
* Written informed consent

Key Exclusion Criteria:

* ECOG performance score >2 (patients aged ≥10 years old) OR Lanksy score ≤50% (patients aged <10 years old)
* Stem Cell Transplant patients only: active significant acute GvHD or moderate/severe chronic GvHD requiring immunosuppressive therapy and/or systemic steroids
* Active CNS involvement of disease
* Active hepatitis B, C or HIV infection
* Oxygen saturation ≤90% on air
* Bilirubin >3 x upper limit of normal
* GFR <30 ml/min
* Cardiac dysfunction
* Patients receiving corticosteroids at a supraphysiological dose that cannot be discontinued
* Known allergy to any component of the ATIMP
* Any contraindications to lymphodepletion or to the use of cyclophosphamide or fludarabine as per local SmPC
* Women who are pregnant or breastfeeding
* Life expectancy <3 months
* Fulminant or rapidly progressive disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2042-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of generation of CARCCR9 T cells as evaluated by the number of therapeutic products generated. | 2 years
  To determine the feasibility of semi-automated autologous CARCCR9 T cells manufacture in patients with r/r T-ALL/T-LBL, in the setting of a Phase I trial.
Incidence of treatment-related adverse events (safety and tolerability) | From CAR T cells infusion until 28 days post infusion
  Incidence of grade 3-5 toxicity causally related to the ATIMP.

SECONDARY OUTCOMES:
Persistence of CARCCR9 T cells | From CAR T cells infusion until 2 years post infusion
  Persistence of circulating CARCCR9 T cells in peripheral blood
Expansion of CARCCR9 T cells | From CAR T cells infusion until 2 years post infusion
  Frequency of circulating CARCCR9 T cells in peripheral blood
Potential efficacy of CARCCR9 T cells | At 1 and 2 years post CAR T cells infusion
  Proportion of responders
Potential efficacy of CARCCR9 T cells | At 1 and 2 years post CAR T cells infusion
  Depth of response
Time to disease progression | From CAR T cells infusion (Day 0) until the date of first documented progression, assessed up to 15 years post CAR T cells infusion.
  Length of time from CAR T cells infusion until disease progression
Event free survival | From CAR T cells infusion (Day 0) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 years post CAR T cells infusion.
  Length of time after a patient receives the CAR T cells and remain free from disease progression, recurrence, or death from any cause.
Overall survival | From CAR T cells infusion (Day 0) until the date of death from any cause, assessed up to 15 years post CAR T cells infusion.
  Length of time from the CAR T cells infusion until death, regardless of the cause

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospitals, London, United Kingdom